CLINICAL TRIAL: NCT02848053
Title: The Long-term Effect of Tianqi Capsule Interventions to Prevent Diabetes in the REDUCES Study: a 8-year Follow-up Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Hubei College of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Lian-fengmei, Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Other Study IDs: REDUCES-01
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Impaired Glucose Tolerance; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Tianqi group: used Tianqi Capsule in the REDUCES study
  Interventions: Other: no intervention
- Placebo group: used placebo in the REDUCES study
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
Objectives: This study is aimed to assess whether Tianqi Capsule interventions have a long-term effect on the risk of diabetes and provide evidence that early intervention by traditional Chinese medicine could delay the progression from impaired glucose tolerance to diabetes.

Study contents: 1.420 participants were followed up for 8 years to assess the long-term effect of Tianqi Capsule. Phone-call followed up was applied to investigate the status of impaired glucose tolerance and orthoglycemic survivors until the end of REDUCES study. 2.To participants that determined the status of glucose metabolism, a variety of ways were used to find the evidence of diagnosis of glucose metabolic status, such as glycemia laboratory sheets from normal hospitals, medical records, the use of antidiabetic drugs or insulin injection, etc. 3. To participants that undiagnosed the status of glucose metabolism, oral glucose tolerance test, blood pressure, weight and blood biochemical analysis were performed to assess the state of glucose metabolism. 4. Questionnaires were given to all the participants to investigate their condition of treatment, diet, exercise and other lifestyle.

DETAILED DESCRIPTION:
Study design: Perspective study Study drug: Tianqi CapsuleInclusion criteria: 1. Subjects have participated in the REDUCES study before; 2. Informed consent forms were needed to participants performed to blood test; 3. Laboratory sheets could be voluntary acquirement by participants that determined the status of glucose metabolism; 4.Subjects were not disabled, and could take care of themselves. 5. Subjects did not suffer the infectious disease.

Exclusion criteria: 1. Subjects did not participate the REDUCES study; 2. Subjects suffered serious mental illness; 3. Subjects suffered severe mental or cognitive impairment; 4. Subjects had a history of drug or alcohol dependence; 5. Subjects have participated in other drug clinical trials in the past 1 month.

Main outcome index: Incidence of diabetes. Secondary outcome index: Body mass index, fasting blood-glucose, postprandial blood sugar, blood lipids, blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have participated in the REDUCES study before;
* Informed consent forms were needed to participants performed to blood test;
* Laboratory sheets could be voluntary acquirement by participants that determined the status of glucose metabolism;
* Subjects were not disabled, and could take care of themselves. 5. Subjects did not suffer the infectious disease.

Exclusion Criteria:

* Subjects did not participate the REDUCES study;
* Subjects suffered serious mental illness;
* Subjects suffered severe mental or cognitive impairment;
* Subjects had a history of drug or alcohol dependence;
* Subjects have participated in other drug clinical trials in the past 1 month.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 420 cases
Sampling Method: Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of diabetes | 0 week

SECONDARY OUTCOMES:
Number of participants with abnormal body mass index values (in kg/m^2) | 0 week
Number of participants with abnormal Triglycerides values (in mmol/L) | 0 week
Number of participants with abnormal Cholesterol values (in mmol/L) | 0 week
Number of participants with abnormal Low density lipoprotein values (in mmol/L) | 0 week
Number of participants with abnormal High density lipoprotein values (in mmol/L) | 0 week
Number of participants with abnormal Systolic Blood Pressure values (in mmHg) | 0 week
Number of participants with abnormal Diastolic Blood Pressure values (in mmHg) | 0 week
Number of participants with abnormal blood glucose values (in mmol/L) | 0 week

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin Tong, PHD, Study Chair — Guang'anmen Hospital of China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lian F, Li G, Chen X, Wang X, Piao C, Wang J, Hong Y, Ba Z, Wu S, Zhou X, Lang J, Liu Y, Zhang R, Hao J, Zhu Z, Li H, Fang Liu H, Cao A, Yan Z, An Y, Bai Y, Wang Q, Zhen Z, Yu C, Wang CZ, Yuan CS, Tong X. Chinese herbal medicine Tianqi reduces progression from impaired glucose tolerance to diabetes: a double-blind, randomized, placebo-controlled, multicenter trial. J Clin Endocrinol Metab. 2014 Feb;99(2):648-55. doi: 10.1210/jc.2013-3276. Epub 2014 Jan 16. PMID 24432995
- Available data/document: Clinical Study Report — http://www.ncbi.nlm.nih.gov/pubmed/?term=Chinese+Herbal+Medicine+Tianqi+Reduces+Progression+From+Impaired+Glucose+Tolerance+to+Diabetes%3A+A+Double-Blind%2C+Randomized%2C+Placebo-Controlled%2C+Multicenter+Trial — This is the original study, the registration study is the follow-up study aimed at Tianqi capsule